CLINICAL TRIAL: NCT01182714
Title: A Prospective Randomized Trial to Compare Immediate and 24-hours Delayed Catheter Removal Following Total Abdominal Hysterectomy
Brief Title: A Prospective Randomized Control Trial Comparing Immediate and 24-hours Delayed Catheter Removal Following Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Dr Joyce Chai, Queen Mary Hospital, University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Foley-01
Record Dates: First submitted 2010-08-11; First posted 2010-08-17 (Estimated); Last update posted 2010-08-20 (Estimated); Status verified 2010-08

CONDITIONS: Hysterectomy
Keywords: Hysterectomy; Catheterisation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- removal of catheter (Other)
  Interventions: Procedure: immediate removal of in-dwelling catheter; Procedure: 24 hours delayed removal of catheter

INTERVENTIONS:
Procedure: immediate removal of in-dwelling catheter
Procedure: 24 hours delayed removal of catheter

SUMMARY:
Total abdominal hysterectomy is a common gynaecological operation performed worldwide. In Hong Kong, it was the most common gynaecological open procedure done and the number of hysterectomies performed increased by almost 50% in 2004 when compared to 1999. In-dwelling catheter use after uncomplicated abdominal hysterectomy has been the standard method for bladder treatment after the operation. It is traditionally advocated to assess urinary output and to prevent post-operative urinary retention as patients with abdominal wound are unable to increase the intra-abdominal pressure to aid voiding. However, in-dwelling catheters have been associated with increased white cell counts and higher rates of positive urine cultures, and subsequently urinary tract infection can lead to increased morbidity, duration of hospital stay, and overall healthcare cost.

Duration of catheter use post-operatively is generally based on custom rather than evidence-based knowledge and therefore varies considerably. The current practice of the investigators hospital is to leave an in-dwelling catheter in-situ for 24 hours after an uncomplicated open gynaecological surgery. Schiotz et al showed that twenty-four-hour catheterization after common gynaecological procedures was associated with a low rate of voiding problems after catheter removal. Post-operative urinary retention leading to bladder atony may increase the long-term morbidity through increased risk of infection, detrusor instability and voiding difficulties. In-dwelling catheter in the immediate post-operative period will help to combat this problem. However, this has to be balanced against the potential risk of catheter-associated urinary tract infection which varies from 5% to 43% in the published trials.

A prospective randomized study comparing immediate versus delayed catheter removal following hysterectomy showed that delayed removal after operation was not associated with an increased rate of febrile events or urinary tract infections, but a significantly higher subjective pain assessment. The size of the catheter used was 16F which was not the standard 12F that the investigators used in the investigators hospital setting. It is postulated that if a smaller caliber in-dwelling catheter is used, it will not result in an increased subjective pain assessment, and the catheter can be left in-situ for 24 hours without causing increased adverse outcomes but possibly reducing recatheterisation rate post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* All women required total abdominal hysterectomy +/- bilateral salpingo-oophorectomy for various benign gynaecological diseases in Queen Mary Hospital

Exclusion Criteria:

* a known history of neurological disorder
* a known history of urinary incontinence
* women who had recurrent urinary tract infections or positive urine culture (>105 colony-forming units of an identified single uro-pathogen per milliliter of urine) pre-operatively
* women for whom a complicated procedure was encountered during the hysterectomy in which case in-dwelling catheter had to be kept post-operatively at the surgeon's decision
* women who had spinal anaesthesia as the choice of anaesthesia or received patient-controlled analgesia as post-operative pain relief.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2007-11; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
the subjective pain assessment provided by the patient post-operatively | post operatively day 1
  pain assessment using visual analogue scale

SECONDARY OUTCOMES:
the rate of recatheterisation | at 6 hours post-operatively
incidence of symptomatic urinary tract infection | up to 7 days after operation

CONTACTS AND LOCATIONS:
Overall Officials: Joyce Chai, MBChB, Principal Investigator — Queen Mary Hospital, University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Ellahi A, Stewart F, Kidd EA, Griffiths R, Fernandez R, Omar MI. Strategies for the removal of short-term indwelling urethral catheters in adults. Cochrane Database Syst Rev. 2021 Jun 29;6(6):CD004011. doi: 10.1002/14651858.CD004011.pub4. PMID 34184246